CLINICAL TRIAL: NCT07011394
Title: Diagnosing Asthma With Clinically Accessible, Non-invasive, and Efficient Tests: a Child-inclusive Translational Investigation
Acronym: DIVE 2
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Association Pulmonaire du Quebec (Other); Fonds de la Recherche en Santé du Québec (Other Government); Fondation JA DeSève (Unknown); Opération Enfant Soleil (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-5346
Record Dates: First submitted 2025-04-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-02

CONDITIONS: Diagnosis; Inflammation; Asthma in Children; Asthma
Keywords: observationnal study; asthma diagnosis; FeNO and eosinophil blood count; children
MeSH Terms: conditions — Disease; Inflammation; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, serum, nasal epithelial lining fluid by nasosorption, urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients aged 6-18 with suspected asthma, referred by primary care for methacholine BPT: Patients will be recruited from a larger study, Propulsion Santé, which investigates the usefulness of FeNO and BEC in prioritizing patients whith suspected asthma for bronchial provocation testing in primary care. 1,500 participants will be invited to receive spirometry at 3 centers: CHUS, CHUSJ, and Montreal Children's Hospital. If spirometry is non-diagnostic, patients aged 6 to 18 years who are referred for methacholine challenge testing will be offered the opportunity to participate in the DIVE2 study.In addition to a medical assessment and standardized questionnaires (ACQ5, ACT, and EQ-5D), participants will undergo FeNO and BEC measurements, and additional blood tests (complete blood count with differential, C-reactive protein, total and specific serum immunoglobulin E, and biobank sample collection). a nasosorption and urine analysis will be performed as part of this protocol.
  Interventions: Diagnostic Test: FeNO; Diagnostic Test: Blood eosinophil count

INTERVENTIONS:
Diagnostic Test: FeNO — FeNO will be measured before the bronchial provocation test using a FeNO VIOX device
Diagnostic Test: Blood eosinophil count — a blood test will be performed om the day of bronchial provocation test

SUMMARY:
Asthma is a common inflammatory respiratory disease affecting 11% of Canadians, but its diagnosis remains challenging, leading to delays in treatment or overtreatment. Spirometry with a reversibility test and bronchial provocation testing (BPT), considered the gold standard, are the reference diagnostic methods. However, access to BPT is limited as it is performed in hospital settings.

Type 2 inflammation biomarkers, the fractional exhaled nitric oxide (FeNO) and blood eosinophils (EOS), represent a potential alternative. In addition to their prognostic and theragnostic value, these markers predict a good response to inhaled corticosteroids in individuals aged ≥ 6 years with asthma. However, their use remains restricted to pulmonologists in specialized clinics and is not recommended as a diagnostic tool in Quebec.

Despite studies demonstrating their diagnostic value in specialized settings, these tests remain underexplored in primary care and insufficiently studied in children under 12 years.

The objective of ou study is to evaluate the relevance and performance of FeNO and blood eosinophils in the diagnosis of asthma in children referred in primary care with non-diagnostic spirometry.

DETAILED DESCRIPTION:
Background Asthma is a common inflammatory airway disease affecting 11% of Canadians. However, its diagnosis remains a significant challenge Spirometry is the first-line diagnostic test, aimed at detecting reversible bronchial obstruction. However, this test yields false-negative results in 40% of cases. The gold standard for diagnosis is the bronchial provocation test; in fact, 80% of patients with a positive provocation test had a normal spirometry result. However, this test requires a lengthy procedure and must be conducted in a hospital setting, making access difficult. Consequently, this leads to both over- and underdiagnosis.

Thus, it is necessary to explore other effective diagnostic methods. Fractional exhaled nitric oxide (FeNO) and blood eosinophil count (BEC) are biomarkers of type 2 inflammation in asthma. Elevated levels are associated with a worse prognosis but also predict a better response to inhaled corticosteroids. These biomarkers have demonstrated diagnostic utility in specialized contexts. However they remain rarely used and lack validation in primary care in Canada, especially in children under 12.

Hypothesis Measuring blood eosinophils and FeNO is a practical and precise diagnostic strategy for children with suspected asthma in primary care when spirometry results are inconclusive.

Objectives This prospective observational study aims to estimate and validate the diagnostic performance of type 2 inflammatory biomarkers, FeNO and/or BEC, in children aged 6 to <18 years referred by primary care providers for suspected asthma with inconclusive pre- and post-bronchodilator spirometry. Additionally, an exploratory analysis will assess inflammatory proteins (alarmins, type 2 cytokines, and chemokines) in serum and nasal epithelial fluid. These objectives will contribute to improving our knowledge of the mechanistic and operational value of type 2 inflammatory biomarkers in an under-studied population.

Methods In parallel with the DIVE study (NCT05992519; Nagano #2023-4791), the investigators propose extending the research to pediatric populations through this twin study (DIVE2), which involves 123 participants aged 6 to <18 years with non-diagnostic pre- and post-bronchodilator spirometry, referred from primary care for bronchial provocation testing. Before this test, participants will have their FeNO measured, undergo a blood test (for BEC, allergy testing, and inflammatory proteins), and nasosorption will be performed. The target sample size of 123 is powered at 90% to calculate the area under the curve (AUC) for three receiver operating characteristic (ROC) curves, with an AUC ≥ 0.7, which is significantly different from the null hypothesis (AUC = 0.5), using a conservatively corrected two-sided α error of < 0.016, assuming a positive/negative case ratio of 2.

These ROC curves will be developed based on the gold standard, bronchial provocation with methacholine (dose causing a 20% drop in FEV1 (DP20) <400 mcg. In line with our institutional procedures, the investigators will not apply the European DP20 threshold of ≤200 mcg but will analyze the impact of other thresholds.

Outcomes :

The primary analysis will assess the diagnostic performance of these biomarkers by calculating the ROC and AUC for FeNO, EOS, and their combination.

The exploratory outcomes are:

* Evaluation of the effectiveness of biomarkers as a diagnostic tool based on diagnostic delay and costs compared to methacholine challenges
* Analysis of biomarker levels in asthmatic patients at the time of diagnosis according to the ORACLE model, for stratification (https://www.oraclescore.com/fr)
* Univariate and multivariate modelling between eosinophils, FeNO, and inflammatory proteins in serum and nasal epithelial fluid (alarmins Thymic stromal lymphopoetin (TSLP) and IL-33; type-2 cytokines IL-4, -5, -13; chemokines eotaxin-3 and thymus activating regulatory cytokine (TARC), prostaglandine-D2 (PGD2), leukotriene-E4 (LTE4), interféron-gamma, tumour necrosis factor alpha (TNF-α))
* Evaluation of participants' and referring physicians' perception of biomarker measurement in relation to asthma diagnosis.
* Longitudinal follow-up of participants to assess medication, symptoms, quality of life, and exacerbations.
* The environmental impact of diagnostic delays due to unnecessary inhaler prescriptions and usage.

Feasibility The University Hospital Centre of Sherbrooke (CHUS), University Hospital Centre of Sainte Justine (CHUSJ), and Montreal Children's Hospital have a waiting list of over 1,300 methacholine challenge tests requested by primary care providers for pediatric patients.

Expected Results: the investigators expect to show type 2 biomarkers such as FeNO and BEC are a practical and effective alternative for diagnosing asthma in primary care particularly when access to standard tests is limited. The investigators expect to strengthen the mechanistic understanding of type 2 inflammatory asthma.

Impact: The investigators aim to provide scientific evidence that biomarkers such as FeNO and blood eosinophils can enhance and accelerate the diagnostic process for children aged 6 to <18 years. Due to their mechanistic, prognostic, and theranostic value, early detection of these biomarkers will allow for the timely initiation of appropriate treatment, ultimately improving asthma management, particularly in the pediatric population. This approach is expected to positively impact the reduction of overdiagnosis and underdiagnosis, benefiting prognosis, quality of life, and offering economic and ecological advantages.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 6 to <18 years, presenting symptoms suggestive of asthma
* Patients referred for a methacholine bronchial provocation test by primary care (defined as non-pulmonologist, non-ENT specialist, non-allergist)
* Spirometry inconclusive

Exclusion Criteria:

* Use of an inhaled or systemic corticosteroid in the previous 48 hours;
* Smoking in the previous 6 hours; history of viral and/or bacterial respiratory infection in the past 4 weeks;
* major cardiopulmonary disease, including: a) chronic obstructive pulmonary disease (COPD), defined by all of the following: i) aged ≥ 40 years , ii) permanent obstruction on spirometry (FEV1/FVC <0.7) and iii) a smoking history of >10 pack-years or known alpha-1-antitrypsin deficiency, b) lung conditions deemed significant by the investigator, including cystic fibrosis and bronchiectasis, and c) unstable heart disease.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be recruited in through two pathways in 3 centers (CHUS, CHUSJ, and Montreal Children's Hospital)
  1. In collaboration with the respiratory physiology department of participating centers, patients scheduled for a methacholine challenge test will receive an invitation letter for the study along with their test appointment notice. They will be informed about the study's purpose, procedures, and provided with contact details to reach out to the research team if they wish to decline participation or have any questions. If no refusal is received, the clinical inhalation therapist will contact them to confirm their eligibility.
  2. Through the Propulsion Santé study, patients will be scheduled for their respiratory test, which will include eosinophil count and FeNO measurement. If their spirometry results are inconclusive for diagnosis, they will be offered the opportunity to participate in the DIVE2 study.
Sampling Method: Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Fractional exhaled nitric oxide value: AUC of the ROC analysis to diagnose asthma | FeNO measured on the day of the methacholine challenge (i.e. Baseline visit)
  Diagnosis of asthma defined as a methacholine PD20 < 200 mcg
Blood eosinophil count value : ROC analysis AUC to diagnose asthma | Blood eosinophils measured on the day of the methacholine challenge (i.e. Baseline visit)
  Diagnosis of asthma defined as a methacholine PD20 < 200 mcg
Combination of FeNO + Blood eosinophil count: ROC analysis AUC to diagnose asthma | Time Frame: FeNO and blood eosinophils measured on the day of the methacholine challenge (i.e. Baseline visit)
  Diagnosis of asthma defined as a methacholine PD20 < 200 mcg

SECONDARY OUTCOMES:
Univariate association between biomarkers (blood eosinophils and FeNO) and inflammatory proteins/metabolites (interleukines, chimiokines, alarmins) | Baseline
  concentration of inflammatory proteins/metabolites (interleukine (IL)-4, IL-5, IL-13, thymic stromal lymphopoietin, leukotriene 4, prostaglandine 2) measured in the NELF, serum analyzed according to FeNO and BEC, and the diagnostic. Further exploratory multivariate modelling adjusting for atopy (defined as a history of eczema, rhinoconjunctivitis, or food allergy and/or at least one sensitisation to an airbourne sensitiser) and biological sex.
Biomarker level in asthmatic patients at time of diagnosis | Baseline
  Expressed as n (%) of diagnosed patients per square in a 3×3 grid stratified by combination of biomarkers (eosinophils <0.15, 0.015-<0.30, ≥0.30×109/L; FeNO <25, 25-<50, ≥50 ppb)
Change in diagnostic delay in asthma patients | Baseline
  the difference (in days) between the date of the non-diagnostic spirometry and the date of the metacholine challenge test
Cost difference between diagnostic strategies | Baseline
  Difference in cost (in Canadian dollars) between the use of biomarkers (FeNO and eosinophil count - analysed separately for traditional vs. point-of-care testing) and the standard methacholine challenge as a second diagnostic step.
Ecological footprint of asthma diagnostic delay | Baseline
  Carbon footprint (in kg CO₂e - carbon dioxide equivalent, as defined by CASCADES Canada) associated with the prescription and use of inhalers prior to the confirmed asthma diagnosis, in the year preceding the methacholine challenge test.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data of this study may be shared if the investigators proposed use of the data has been approved by the study principal investigator and an institutional research ethics committee.
Access Criteria: Data of this study may be shared if the investigators proposed use of the data has been approved by the study principal investigator and an institutional research ethics committee.

REFERENCES:
- [Derived] Gronnier M, Desy L, Pouliot L, Lemieux SE, Vezina FA, Lachapelle P, Counil FP, Duval M, Cliche D, Lemaire-Paquette S, Coulibaly L, Hudon C, Lands LC, Ducharme FM, Tse S, Couillard S. Integrating blood eosinophils and exhaled nitric oxide (FeNO) in asthma diagnostic pathways for adults and children: the PROPULSION SANTE observational study with translational sub-studies (DIVE, DIVE2)-protocols. BMJ Open Respir Res. 2025 Nov 27;12(1):e003750. doi: 10.1136/bmjresp-2025-003750. PMID 41314665